CLINICAL TRIAL: NCT03027908
Title: A Study to Measure the Effect of Two Fluoride Toothpastes on Gingival Health Over a Six Month Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ORL-GUM-2544
Record Dates: First submitted 2016-12-09; First posted 2017-01-23 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoride Toothpaste 1 (Experimental): Toothpaste containing Sodium Fluoride at 1450 ppm F
  Interventions: Other: Fluoride Toothpaste 1
- Fluoride Toothpaste 2 (Active Comparator): Toothpaste containing Sodium Fluoride at 1450 ppm F
  Interventions: Other: Fluoride Toothpaste 2

INTERVENTIONS:
Other: Fluoride Toothpaste 1 — Toothpaste containing 1450 ppm F as Sodium Fluoride
  Other Names: A1
  Arms: Fluoride Toothpaste 1
Other: Fluoride Toothpaste 2 — Toothpaste containing 1450 ppm F as Sodium Fluoride
  Other Names: A2
  Arms: Fluoride Toothpaste 2

SUMMARY:
This study is a double-blind, randomised, parallel group efficacy study. A minimum of 240 healthy female and male participants aged over 18 years will participate. The participants will be randomised into two groups. Participants will be randomly assigned to the test groups according the allocation table prepared by the Statistician.

Participants will be enrolled on to the study according to the inclusion/exclusion criteria. After enrollment participants will have their teeth cleaned using a professional prophylaxis polish by the study hygienist. The participants will then be provided with a standard cosmetic silica fluoride toothpaste and a toothbrush to use at home, twice a day for up to four weeks. After this time, they will return to the test site and have the baseline dental assessments. Participants will then be randomly allocated to one of the two test products which they will use at home, twice a day for the duration of the study. Dental assessments will be conducted after 13 and 26 weeks of product use at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and physically able to carry out all study procedures.
* Be willing and competent (verbally and cognitively) to give written informed consent and complete a medical history form.
* Have at least 20 natural teeth including 5 teeth (excluding 3rd molars) in each quadrant
* Have a mean Modified Gingival Index (MGI) score of between 2.00 and 2.75 at screening.
* Not have had a scale and prophylaxis in the month prior to enrolment or have one scheduled prior to the end of the study.
* Be willing to use only the test products for 6 months

Exclusion Criteria:

* Current participation in any other cosmetic trials, any dental clinical trials or clinical trials.
* Pregnant or breast feeding mothers.
* Medical condition and/or regular use of any medication which might affect the outcome of the study, as determined by the study dentist, principally a course of anti-inflammatory, antimicrobial or statin drugs
* Obvious signs of untreated caries or significant periodontal disease, which in the opinion of the Study Dentist, will affect either the scientific validity of the study or if the participant was to participate in the study would affect their wellbeing.
* Any participant who, in the judgement of the investigator, should not participate in the study.
* Full or partial dentures wearers.
* Current orthodontic treatment.
* Have oral piercings.
* Smokers or those who have a recent smoking history, including e-cigarettes.
* Taking dietary supplements (e.g. multivitamins; antioxidants; fish oils).
* Any subject with a single MGI score of 4 in the any area of the mouth at any time point will be excluded.
* A subject will be excluded from the study if they have a MGI mouth mean of greater than 2.75 at screening
* Any subject with a single MGI score of 3 at Baseline
* Use of non study oral care products, e.g. dental floss, chewing gum, mouth rinses during the pre treatment and test phases of the study.
* The subject is an employee of Unilever or a member of the study team.
* Taking a course of antimicrobial or anti-inflammatory drugs within 4 weeks of screening
* Those taking anti-histamine or anti-inflammatory medication in the 24 hours prior to the dental assessments
* Diabetics
* Vegetarians and Vegans

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Change in gingival condition as measured by the Modified Lobene Gingival Index | 13 weeks
Change in gingival condition as measured by the Saxton van der Ouderaa bleeding index | 13 weeks
Change in plaque levels as measure by the Quigley and Hein Plaque index | 13 weeks

SECONDARY OUTCOMES:
change in gingival condition as measured by the Modified Lobene Gingival Index | 26 weeks
change in gingival condition as measured by the Saxton van der Ouderaa bleeding index | 26 weeks
Change in plaque levels as measured by the Quigley and Hein plaque index | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola X West, Professor, Principal Investigator — University of Bristol

IPD SHARING:
Plan to Share IPD: No